CLINICAL TRIAL: NCT00212069
Title: Serum Protein Profiling as a Predictor of Gemcitabine Sensitivity in Breast Cancer With Prior Exposure to Anthracyclines and Taxanes
Brief Title: Serum Proteomics to Predict Gemcitabine Sensitivity in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR01/12/03
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; serum proteomics; gemcitabine; carboplatin; chemotherapy sensitivity
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Carboplatin

INTERVENTIONS:
Drug: gemcitabine, carboplatin

SUMMARY:
Tumors are heterogeneous with varying response to chemotherapeutic agents. We hypothesize that tumors that are sensitive to a particular chemotherapeutic agent have a distinctive tumor protein profile compared to those that are resistant. We further hypothesize that since tumor is continuously perfused by serum, serum protein profile can be used as a surrogate marker of tumor protein profile. The primary objective of this study is to identify a serum protein profile that predicts gemcitabine/carboplatin sensitivity or resistance in breast cancer patients with prior exposure to anthracyclines and taxanes. Secondary objectives are to establish the serum protein profile of breast cancer patients who have had prior exposure to anthracyclines and taxanes, and to study the pharmacogenetics of gemcitabine toxicity by correlating germline genotype of transporters and drug metabolizing enzymes with plasma and intracellular gemcitabine pharmacokinetics.

DETAILED DESCRIPTION:
Metastatic breast cancer patients previously treated with anthracyclines and taxanes will be treated with gemcitabine and carboplatin every 3 weeks. Serial plasma samples will be collected for proteomics profiling with SELDI-MS that will be correlated with tumor response to identify biomarkers that may predict for chemotherapy sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Female, age >= 18 years.
* Histologic or cytologic diagnosis of breast carcinoma.
* Stage IV breast cancer with prior exposure to anthracyclines and taxanes, either in the neoadjuvant, adjuvant or metastatic setting.
* Presence of at least one uni-dimensionally measurable, non-CNS indicator lesion defined by radiologic study or physical examination
* For patients with previous radiotherapy, the indicator lesion(s) must not be within the previous radiation field. The last dose of radiotherapy should be at least 3 weeks prior to study entry. The total radiotherapy received should not be more than 30% of the bone marrow.
* Karnofsky performance status of 70 or higher.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  - Bone marrow: White blood cells (WBC) >= 3.5 x 109/L Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 109/L Platelets >= 100 x 109/L Haemoglobin >= 9g/dL

  - Hepatic: Bilirubin <= 1.5 x upper limit of normal (ULN), ALT or AST <= 2.5x ULN, (or <5 X with liver metastases) Alkaline phosphatase <= 2.5x ULN.

  - Renal: Creatinine clearance >30ml/minute, based on the Cockcroft formula
* Signed informed consent from patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-03; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To identify a serum protein profile that predicts gemcitabine/carboplatin sensitivity or resistance in breast cancer patients with prior exposure to anthracyclines and taxanes.

SECONDARY OUTCOMES:
a. To establish the serum protein profile of breast cancer patients who have had prior exposure to anthracyclines and taxanes.
b. To study the pharmacogenetics of gemcitabine toxicity by correlating germline genotype of transporters and drug metabolizing enzymes with plasma and intracellular gemcitabine pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Chin Lee, MD, Principal Investigator — Consultant
Locations (1):
- National University Hospital, Singapore, Singapore